CLINICAL TRIAL: NCT05784506
Title: Metabolites Profiling Reveals Nutrient Processing Patterns Upon Dietary Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yang Tao, Professor, Chief physician, Nanjing Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-SR-298
Record Dates: First submitted 2023-02-20; First posted 2023-03-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Metabolism Disorder; Nutrition
MeSH Terms: conditions — Metabolic Diseases | interventions — Nutrients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Macronutrients loading test for healthy group (Experimental): A total of 30 subjects with normal metabolic status underwent four successive food tolerance tests (glucose, protein, butter and olive oil) at one-week intervals.
  Interventions: Other: Macronutrients
- Mixed meal tolerance test (MMTT) for healthy group (Experimental): A total of 40 subjects with normal weight and plasma glucose levels underwent MMTT.
  Interventions: Other: Mixed meal tolerance test (MMTT)
- Mixed meal tolerance test (MMTT) for overweight subjects with normal plasma glucose (Experimental): A total of 40 overweight subjects without a history of diabetes underwent MMTT.
  Interventions: Other: Mixed meal tolerance test (MMTT)
- Mixed meal tolerance test (MMTT) for obese subjects with abnormal plasma glucose (Experimental): A total of 40 obese subjects without a history of diabetes underwent MMTT.
  Interventions: Other: Mixed meal tolerance test (MMTT)

INTERVENTIONS:
Other: Macronutrients — Four successive food tolerance tests (glucose, protein, butter and olive oil) at one-week intervals.
  Arms: Macronutrients loading test for healthy group
Other: Mixed meal tolerance test (MMTT) — Mixed meal tolerance test (MMTT)
  Arms: Mixed meal tolerance test (MMTT) for healthy group; Mixed meal tolerance test (MMTT) for obese subjects with abnormal plasma glucose; Mixed meal tolerance test (MMTT) for overweight subjects with normal plasma glucose

SUMMARY:
The reasonable combination of macronutrients including carbohydrates, proteins and fat, is the basis of rational diet and beneficial to treatment of metabolic diseases including obesity and diabetes. Endocrine hormones play pivotal roles in regulation of nutrients metabolism and energy homeostasis. However, the dynamic metabolism following the consumption of macronutrients and the relationship between various metabolites and endocrine hormones during these procedures yet to be adequately explained nowadays. Therefore, in this study, the investigators selected glucose, protein, fat and mixed meal tolerance test (MMTT) for the loading tests, endocrine hormones and metabolites were detected to profile the molecular changes in the plasma. The investigators aimed to explore the nutrient processing patterns of various macronutrients and determine the interaction between metabolic hormones and metabolites.

ELIGIBILITY:
Inclusion Criteria:

1. Those who agree to participate in the study and sign informed consent.
2. Age between 20 and 65 year.
3. Fasting plasma glucose < 7.0mmol/l, and 2-hour postprandial plasma glucose < 11.1mmol/l.
4. BMI > 18 kg/m2.

Exclusion Criteria:

1. History of diabetes.
2. Pregnant or lactating women.
3. The subjects had not received oral/systemic corticosteroids for 7 consecutive days during the last 6 months.
4. Subjects were taking medication known to affect glucose metabolism.
5. Subjects who take strong inhibitors of cytochrome P450 (CYP)3A4/5, for example, ketoconazole, azanaway, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir and telithromycin.
6. Patients with either of the following characteristics of severe hepatic disease:

   i. Two consecutive abnormal hepatic function results during recent four weeks, with ALT or AST three times the upper limit of the institutions normal reference ranges.

   ii. Hepatic excretion dysfunction (eg. hyperbilirubinemia) and/or synthesis dysfunction, or other decompensated liver disease.

   iii. Acute viral hepatitis, autoimmune hepatitis, and alcoholic hepatitis
7. Patients with moderate and severe renal impairment, and end-stage renal disease (serum creatinine > 194.5 mmol/L, or serum potassium > 5.5 mmol/L).
8. New York Heart Association (NYHA) functional class III or IV congestive heart failure.
9. History of acute or chronic pancreatitis.
10. History of gastrointestinal disorders: gastroenterostomy, enterectomy, ileus and intestinal ulcers.
11. Subjects with previously diagnosed malignancy within the past 5 years.
12. Any other reasons that the investigator considered inappropriate to participate in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Metabolites | 0 to 180 minutes after a dietary loading
  Plasma metabolites after dietary loading.
Endocrine hormones | 0 to 180 minutes after a dietary loading
  Plasma insulin and C-peptide after dietary loading.
Proteomics | 0 to 180 minutes after a dietary loading
  Plasma proteomics after dietary loading.
Lipidomics | 0 to 180 minutes after a dietary loading
  Plasma lipidomics after dietary loading.
Diet questionnaire | 3 days
  Diet questionnaire
Stool microbiome | Baseline
  Metagenomic sequencing and 16s microbiome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, MD/PhD, Study Chair — First Affiliated Hospital, Nanjing Medical University
Locations (1):
- First Affiliated Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

DOCUMENTS (1):
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT05784506/ICF_000.pdf